CLINICAL TRIAL: NCT03179215
Title: Dynamic Arterial Elastance as a Predictor of Arterial Blood Pressure Response to Fluid Administration in Septic Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, soudy salah hammad, Anesthesia, ICU and pain management assistant lecturer ,Aswan University, Cairo University
Other Study IDs: N-35 -2017
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: fluid challange — A set of hemodynamic measurements will be obtained at baseline and after infusing a fluid challenge (FC) of 150-250 ml normal saline over 5-10 minutes.Fluid-responders are patients with a SV increase ≥10% after fluid challenge

SUMMARY:
Correction of arterial hypotension is essential for adequate cellular metabolism. maintaining MAP above a minimum level has been recommended in order to prevent further tissue hypoperfusion and organ dysfunction.Functional assessment of arterial load by dynamic arterial elastance (Eadyn), has recently been shown to predict the arterial pressure response to volume expansion (VE) in hypotensive, preload-dependent septic patients.

DETAILED DESCRIPTION:
After approval from the ethics and research committee of Faculty of Medicine, Cairo University, an informed consent will be obtained from each patient's next of kin. Arteial cathter will be inserted in radial artery and connected through an arterial line to invasive arterial blood pressure monitor. Electrical Cardiometry will be attached to patient through the placement of four skin sensors on the neck and left side of the thorax12. A set of hemodynamic measurements will be obtained at baseline and after infusing a fluid challenge (FC) of 150-250 ml normal saline over 5-10 minutes.Fluid-responders are patients with a SV increase ≥10% after fluid challenge (FC).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (more than 18 years).
* Sepsis as a cause of admission.

Exclusion Criteria:

* • Patients younger than 18 years of age.

  * Pregnant females.
  * Trauma as a cause of intensive care unit (ICU)admission.
  * Known medical history of vasodilator therapy.
  * Cardiac arrhythmias.
  * Any absolute contraindication for fluid administration such as congestive heart failure, pulmonary edema and/or fluid overload

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients with the diagnosis of sepsis who will be admitted to the Trauma and Surgical Intensive Care Unit (SICU) of Kasralainy School of Medicine,Cairo University during a 6-month period (from March 2017 to September 2017) will be enrolled in the study.Sepsis is defined according to Surviving Sepsis Campaign: International Guidelines for Management of Severe Sepsis and Septic Shock: 2016 as life-threatening organ dysfunction due to a dysregulated host response to infection.10 Septic shock is defined as a subset of sepsis in which particularly profound circulatory, cellular, and metabolic abnormalities substantially increase mortality.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
dynamic arterial elastance | 6 month
  confirm the ability of non invasive (Eadyn) for predicting arterial pressure response to fluid challenge in septic patients

CONTACTS AND LOCATIONS:
Overall Officials: ahmed m mukhtar, proffesor, Principal Investigator — Cairo University
Locations (1):
- Trauma & Surgical ICU. New Emergency Hospital (185 Hospital), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia MI, Romero MG, Cano AG, Aya HD, Rhodes A, Grounds RM, Cecconi M. Dynamic arterial elastance as a predictor of arterial pressure response to fluid administration: a validation study. Crit Care. 2014 Nov 19;18(6):626. doi: 10.1186/s13054-014-0626-6. PMID 25407570
- [Background] Cecconi M, Monge Garcia MI, Gracia Romero M, Mellinghoff J, Caliandro F, Grounds RM, Rhodes A. The use of pulse pressure variation and stroke volume variation in spontaneously breathing patients to assess dynamic arterial elastance and to predict arterial pressure response to fluid administration. Anesth Analg. 2015 Jan;120(1):76-84. doi: 10.1213/ANE.0000000000000442. PMID 25230102